CLINICAL TRIAL: NCT05718570
Title: A Multi-national, Multi-centre, Prospective, Single-arm, Observational, Non-interventional Post-authorisation Safety Study to Investigate Long-term Safety of Sogroya® (Somapacitan) in Adults With Growth Hormone Deficiency (AGHD) Under Routine Clinical Practice
Brief Title: A Study to Follow Patients With Adult Growth Hormone Deficiency (AGHD) Treated With Sogroya® for Long Term Safety Information
Status: Enrolling by invitation | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN8640-4515; U1111-1264-8642 (Other: World Health Organization (WHO))
Record Dates: First submitted 2023-01-30; First posted 2023-02-08 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Adult Growth Hormone Deficiency
MeSH Terms: conditions — Dwarfism, Pituitary | interventions — somapacitan

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with Adult Growth Hormone Deficiency (AGHD): Participants will be treated with commercially available Sogroya according to routine clinical practice at the discretion of the treating physician. The decision to treat a participant with Sogroya has been made prior to and independently from the decision to include the participant in this study.
  Interventions: Drug: Somapacitan

INTERVENTIONS:
Drug: Somapacitan — Sogroya therapy in participants with AGHD.

SUMMARY:
In this study, the general long-term safety and effectiveness of Sogroya (somapacitan) in adults with growth hormone deficiency (AGHD) being treated per normal clinical practice is looked into. In the study, information on side effects and how well Sogroya (somapacitan) works during long term treatment in people with Adult Growth Hormone Deficiency (AGHD) will be collected and analysed. Participants will be treated with Sogroya (somapacitan) as prescribed by the study doctor, in accordance with normal clinical practice. The study will last for 5-10 years, depending on when the participant join the study. The participant will be asked to complete two short questionnaires during every visit to the clinic. The questionnaires will collect information on the participant's well-being, work ability and ability to perform daily activities.

ELIGIBILITY:
Inclusion Criteria:

1. Signed consent obtained before any study-related activities (study-related activities are any procedure related to recording of data according to the protocol).
2. The decision to initiate treatment with commercially available Sogroya (somapacitan) has been made by the participant and the treating physician before and independently from the decision to include the participant in this study.
3. Male or female, age above or equal to 18 years assigned to Sogroya (somapacitan) treatment at the time of signing informed consent.
4. Diagnosis of adult growth hormone deficiency (AGHD) as per local practice.

Exclusion Criteria:

1. Previous participation in this study. Participation is defined as signed informed consent.
2. Mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation.
3. Participant with hypersensitivity to the active substance or to any of the excipients.
4. Participant with active malignancy or in treatment for active pre-existing malignancy.
5. Participant with acute critical illness, suffering from complications following open heart surgery, abdominal surgery, multiple accidental trauma, acute respiratory failure or similar conditions per investigator judgement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with Adult Growth Hormone Deficiency
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-02-03 (Actual); Primary Completion 2032-12-15 (Estimated); Study Completion 2032-12-15 (Estimated)

PRIMARY OUTCOMES:
Number of Adverse drug reaction (ADRs) | From baseline (week 0) to end of study (between 1 week and a maximum of 10 years)
  Measured as count of events.
Incident Neoplasm | From baseline (week 0) to end of study (between 1 week and a maximum of 10 years)
  Measured as number of participants (yes/no).
Incident Diabetes Mellitus type 2 | From baseline (week 0) to end of study (between 1 week and a maximum of 10 years)
  Measured as number of participants (yes/no).

SECONDARY OUTCOMES:
Number of Adverse Events (AEs) | From baseline (week 0) to end of study (between 1 week and a maximum of 10 years)
  Measured as count of events.
Number of Serious Adverse Events (SAEs) | From baseline (week 0) to end of study (between 1 week and a maximum of 10 years)
  Measured as count of events.
Number of Medication Errors (incorrect dose administration rate) | From baseline (week 0) to end of study (between 1 week and a maximum of 10 years)
  Measured as count of errors.
Change in Insulin-like Growth Factor I (IGF-I) standard deviation score (SDS) | From baseline (week 0) to end of study (between 1 week and a maximum of 10 years)
  Measured as score ranging from -10 to +10.
Patient achieving Insulin-like Growth Factor I (IGF-I) standard deviation score (SDS target) (0-+2) | Approximately (closest routine clinical) 12 months after enrolment in study
  Measured as number of participants (yes/no).
Change in Weight | From baseline (week 0) to end of study (between 1 week and a maximum of 10 years)
  Measured as kilogram (kg).
Change in Body Mass Index (BMI) | From baseline (week 0) to end of study (between 1 week and a maximum of 10 years)
  Measured as kilogram per square meter (kg^m2).
Change in waist circumference | From baseline (week 0) to end of study (between 1 week and a maximum of 10 years)
  Measured as centimeter (cm).
Change in waist-hip ratio | From baseline (week 0) to end of study (between 1 week and a maximum of 10 years)
  Measured as ratio.
Change in lipid profile (cholesterol, High Density Lipoprotein [HDL], Low Density Lipoprotein [LDL], triglycerides) | From baseline (week 0) to end of study (between 1 week and a maximum of 10 years)
  Measured as milligrams per deciliter (mg/dL).
Change in glycated hemoglobin (HbA1C) | From baseline (week 0) to end of study (between 1 week and a maximum of 10 years)
  Measured as percentage (%).
Change in bone density | From baseline (week 0) to end of study (between 1 week and a maximum of 10 years)
  Measured as grams per square centimeter (g/cm^2).
Change in bone mineral content | From baseline (week 0) to end of study (between 1 week and a maximum of 10 years)
  Measured as grams (g).
Change in total body fat-mass | From baseline (week 0) to end of study (between 1 week and a maximum of 10 years)
  Measured as kg.
Change in truncal fat-mass | From baseline (week 0) to end of study (between 1 week and a maximum of 10 years)
  Measured as kg.
Change in lean body mass | From baseline (week 0) to end of study (between 1 week and a maximum of 10 years)
  Measured as kg.
Change in body fat percentage | From baseline (week 0) to end of study (between 1 week and a maximum of 10 years)
  Measured as %.
Change in visceral adipose tissue (VAT) | From baseline (week 0) to end of study (between 1 week and a maximum of 10 years)
  Measured as cm^2.
Change in Liver function (Aspartate aminotransferase [AST], Alanine transaminase [ALT], Gamma-Glytamyltransferase [GGT], bilirubin) | From baseline (week 0) to end of study (between 1 week and a maximum of 10 years)
  Measured as Units per liter (U/L).
Change in Patient reported outcome (PRO) score, Treatment Related Impact Measure-Adult Growth Hormone Deficiency (TRIM-AGHD) | From baseline (week 0) to end of study (between 1 week and a maximum of 10 years)
  Measured as score ranging from -100 to +100. Lower score indicates a better health state.
Patient reaching satisfactory clinical response | Approximately (closest routine clinical) 12 months after enrolment in study
  Measured as number of participants (yes/no).

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (55):
- United States (29):
  - Barrow Neurological Institute, Phoenix, Arizona
  - Keck Medical Center of USC - Outpatient Clinic, Los Angeles, California
  - UCLA Health, Los Angeles, California
  - Stanford Univ School of Med, Palo Alto, California
  - Advanced Rx Clinical Research, Westminster, California
  - Anschutz Outpatient Pavilion, Aurora, Colorado
  - Metabolic Research Institute Inc, West Palm Beach, Florida
  - Atlanta Diabetes Associates, Atlanta, Georgia
  - Northwestern Medical Group, Chicago, Illinois
  - Johns Hopkins University, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Washington University, St Louis, Missouri
  - UNMC, Omaha, Nebraska
  - Palm Research Center Inc-Vegas, Las Vegas, Nevada
  - Northern Nevada Endocrinology, Reno, Nevada
  - NYU Langone Health, New York, New York
  - Cornell University, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Physicians East Endocrinology, Greenville, North Carolina
  - Oregon Health & Science University, Portland, Oregon
  - St Lukes Physician Group, Center Valley, Pennsylvania
  - Revival Research Institute, LLC, Dallas, Texas
  - UT Southwestern Medical Center-CRU, Dallas, Texas
  - EP Premier Medical Group PA, El Paso, Texas
  - Consano Clinical Research, LLC, Shavano Park, Texas
  - Puget Sound VA, University of Washington, Seattle, Washington
  - University Of Washington_Seattle, Seattle, Washington
- France (5):
  - HCL - HOPITAL LOUIS PRADEL - Service d'endocrinologie, Bron
  - CHU LILLE - HOPITAL CLAUDE HURIEZ - Service d'endocrinologie et diabétologie, Lille
  - APHM - HOPITAL DE LA CONCEPTION - Service d'endocrinologie, Marseille
  - APHP - LA PITIE SALPETRIERE - Service endrocrinologie et medecine de la reproduction, Paris
  - CHU REIMS - HOPITAL ROBERT DEBRE - Service Endocrinologie-Diabète-Nutrition, Reims
- Germany (10):
  - Uniklinik Aachen - Endokrinologie und Diabetologie, Aachen
  - Endokrinologikum Frankfurt, Frankfurt am Main
  - Universitätsklinikum Halle - Innere Medizin III, Halle
  - Universitätsmedizin der JGU Mainz - Endokrinologie und Stoffwechselerkrankungen, Mainz
  - LMU Klinikum Großhadern München - Med. Klinik, München
  - Medicover Neuroendokrinologie MVZ München, München
  - Medicover Neuroendokrinologie MVZ, München
  - Medicover MVZ Oldenburg, Oldenburg
  - Medicover Oldenburg MVZ, Oldenburg
  - Universitätsklinikum Würzburg - Zentrum für Innere Medizin (ZIM), Würzburg
- Japan (6):
  - Fukuoka University Chikushi Hospital_Endocrinology and Diabetes Mellitus, Chikushino-shi, Fukuoka
  - Kagoshima University Hospital_Neurosurgery, Kagoshima-shi, Kagoshima
  - Nippon Medical School Musashikosugi Hospital_Neurological Surgery, Kawasaki-shi, Kanagawa
  - Kobe University Hospital_Diabetes and Endocrinology, Kobe-shi, Hyogo
  - Okayama University Hospital_General Medicine, Okayama-shi, Okayama
  - Osaka City General Hospital_Endocrinology and Diabetes Mellitus, Osaka-shi, Osaka
- Saudi Arabia (4):
  - Dr Soliman Fakeeh Hospital, Jeddah
  - My clinic, Jeddah
  - Dr. Sulaiman Al Habib Medical Group- Olaya, Riyadh
  - King Fahad Medical City, Riyadh
- UKC Ljubljana, Endocrinology and Diabetes, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com